CLINICAL TRIAL: NCT02971046
Title: Glutathione (GSH) Synthesis in Response to Graded Protein Intakes: a Functional Measure of Protein Requirement in Healthy School-aged Children and Healthy Young and Old Adults
Brief Title: Glutathione (GSH) Synthesis in Healthy School-aged Children and Healthy Young and Old Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Glenda Courtney-Martin, Academic &Clinical Specialist, Project Investigator, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1000053342
Record Dates: First submitted 2016-11-11; First posted 2016-11-22 (Estimated); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Healthy
Keywords: healthy children; protein; glutathione; protein requirement; healthy young adults; healthy adults over 60 years of age

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Protein intake (Experimental): Varying protein intakes.
  Interventions: Other: varying protein intakes

INTERVENTIONS:
Other: varying protein intakes — In healthy school-aged children: Four randomly assigned levels of protein intake in a repeated measured design. The levels of protein intake are 0.95, 1.3,1.55, and 2.0 grams per kilogram of bodyweight per day.
  In healthy young and old adults: Up to six randomly assigned levels of protein intake in a repeated measured design. The levels of protein intake are : 0.66, 0.8, 1, 1.2, and 1.5 grams per kilogram of bodyweight per day.

SUMMARY:
To measure the fractional and absolute synthesis rates of GSH, an antioxidant that protects cells from damage, in the erythrocytes of healthy school-aged children, young adults and old adults in response to graded intakes of protein in order to determine if increasing the protein intake above the current recommended DRI produces increases in the GSH synthesis rates in erythrocytes of these individuals. Participants will consume specially formulated diets with varying protein levels.

DETAILED DESCRIPTION:
The current dietary reference intake (DRI) recommendations for protein in children (6-11 years old) and adults (>19 years old) are based on nitrogen balance data and set at a mean (EAR) of 0.76 and 0.66 g/kg/day respectively and population safe (RDA) recommendation of 0.95 and 0.80 g/kg/day respectively. Using the indicator amino oxidation (IAAO) method we estimated higher protein requirements in these populations. This suggests that current recommendations are underestimated. Studies in adults have shown that protein recommendation set on the basis of nitrogen balance data, while sufficient to maintain nitrogen balance, does not maintain GSH status.

Glutathione (GSH) is most important intracellular antioxidant and scavenger and its deficiency has been shown to compromise recovery in acute as well as chronic stressors. Deficiency of GSH results when protein and/or cysteine intake is inadequate. Inadequate protein intake in children not only compromises growth, but could increase susceptibility to, and compromise recovery from regular childhood illness. Similarly, in young and older adults' inadequate intakes may result in increased oxidative stress and compromised immune function. Measurement of GSH synthesis provides a functional method whereby the current protein recommendation can be tested against higher estimates derived using the IAAO method. The purpose of this study therefore is to measure GSH synthesis in healthy school aged children (6-11 years), and healthy young (19 - 40 years) and old (60 - 90 years) adults in response to current recommended protein intakes and in response to protein requirement estimates derived using the IAAO method.

In healthy school-aged children, each level of protein will be studied over three days. For two days (adaptation days), participants will eat some low protein foods plus a milkshake drink. On the study day, participants will consume 8 hourly protein drinks and special cookies at SickKids. In healthy young and old adults, each level of protein will be studied over three days. For two days (adaptation days), young adults will eat some low protein foods plus a milkshake drink. On the one study day, young adults will consume 10 hourly milkshake diets at SickKids. In old adults, each level of protein will be studied over four days. For three days (adaptation days), old adults will eat some low protein foods plus a milkshake drink. On the one study day, old adults will consume 10 hourly milkshake diets at SickKids.

ELIGIBILITY:
Inclusion Criteria in:

1. Healthy school-aged children

   * Body weight ≥ 22 kg
   * No history of anemia
   * Willingness to participate
2. Healthy Young Adults

   * Consent provided
   * Aged 19 - 40 years old
   * In good general health as evidenced by medical history, physical health and blood draw
   * Fasting blood glucose, hemoglobin A1c (HbA1c), urea, creatinine, vitamin-B6, vitamin-B12 and folate levels within normal ranges for age.
   * Willingness to participate in the study.
   * BMI <25 kg/m2.
3. Healthy Old Adults

   * Consent provided
   * Aged 60- 90 years old
   * In good general health as evidenced by medical history, physical health and blood draw
   * Fasting blood glucose, hemoglobin A1c (HbA1c), urea, creatinine, vitamin-B6, vitamin-B12 and folate levels within normal ranges for age.
   * Willingness to participate in the study.
   * BMI <30 kg/m2.

Exclusion Criteria in:

1. Healthy school-aged children

   * HIV
   * Diabetes
   * Anaemia
   * Significant weight loss within 30 days of study
   * On weight loss diets
   * Body weight less that 22kg
   * Inability to tolerate diet
   * Unwilling to have blood drawn
2. Healthy Young and Old Adults:

   * Presence of chronic disease and/or acute illness known to affect GSH and/or protein/amino acid metabolism (e.g. HIV, diabetes, cancer, liver or kidney disease, acute cold or flu).
   * Anemia (15 - 20% outside lower limit of normal lab reference ranges)
   * Taking medications known to affect GSH and/or protein/AA metabolism (e.g. acetaminophen, steroids).
   * Significant weight loss during the past month or consumption of weight reducing diets.
   * Significant caffeine consumption (>2 cups per day).
   * Significant consumption of alcohol (>1 drink per day i.e. 1 beer or ½ glass of wine).
   * Inability to tolerate the diet
   * Unwilling to have blood drawn from a venous access during the isotope infusion day.

Ages: 6 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Erythrocyte GSH Fractional synthesis rates | up to 24 months
  To measure the fractional synthesis rates of GSH in the erythrocytes of healthy school-aged children and healthy young and old adults in response to graded intakes of protein.

SECONDARY OUTCOMES:
Erythrocyte GSH absolute synthesis | up to 24 months
  To determine the absolute synthesis rate of GSH in erythrocyte of healthy school aged children and healthy young and old adults in response to varying protein intakes.

CONTACTS AND LOCATIONS:
Overall Officials: Glenda Courtney-Martin, PhD, Principal Investigator — Academic &Clinical Specialist
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Paoletti A, Pencharz PB, Rafii M, Tomlinson C, Kong D, Xu L, Elango R, Courtney-Martin G. Protein intake affects erythrocyte glutathione synthesis in healthy adults aged >/=60 years in a repeated-measures trial. Am J Clin Nutr. 2024 Apr;119(4):917-926. doi: 10.1016/j.ajcnut.2024.02.002. Epub 2024 Feb 5. PMID 38325765
- [Derived] Szwiega S, Xu L, Rafii M, Pencharz PB, Kong D, Tomlinson C, Elango R, Courtney-Martin G. Protein intake affects erythrocyte glutathione synthesis in young healthy adults in a repeated-measures trial. Am J Clin Nutr. 2024 Feb;119(2):371-383. doi: 10.1016/j.ajcnut.2023.11.008. Epub 2023 Nov 20. PMID 37992970